CLINICAL TRIAL: NCT06032832
Title: The Effect of Dephytinization on Iron Absorption From a Soy Protein Based Meat Analog, Compared to a Reference Pork Meat Meal: a Randomized Study in Young Women
Brief Title: Iron Absorption From Naturally Dephytinized Legumes
Acronym: LINDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diego Moretti (Other)
Responsible Party: Sponsor-Investigator, Diego Moretti, Prof.Dr. Diego Moretti, Swiss Distance University of Applied Sciences
Organization: Swiss Distance University of Applied Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Iron_LINDA_2023
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Iron Deficiencies
Keywords: plant based meat alternative; iron absorption; soy protein; phytic acid; dephytinization
MeSH Terms: conditions — Iron Deficiencies | interventions — Pork Meat

STUDY DESIGN:
Intervention Model Description: Randomized control trial, cross-over
Who Masked: Participant
Masking Description: Test meals will be randomized and served to participants. Participants will not know or taste the differences of dephytinization in soy protein concentrate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Soy protein concentrate meat analog (Experimental): Meat analog made from soy protein concentrate contains 57Fe as ferrous sulfate. All participants will consume this test meal.
  Interventions: Other: soy protein concentrate-meat analog
- Soy protein concentrate meat analog without phytic acid (Experimental): Meat analog made from soy protein concentrate that was removed phytic acid (dephytinization) contains 58Fe as ferrous sulfate. All participants will consume this test meal.
  Interventions: Other: soy protein concentrate-meat analog_dephytinization
- minced pork meat (Experimental): A meal based on minced pork meat, containing 57Fe intrinsically, will be prepared and served to the participants. All participants will consume this test meal.
  Interventions: Other: pork meat

INTERVENTIONS:
Other: soy protein concentrate-meat analog — Baked Meat analogs-soy protein concentrate containing 57Fe as ferrous sulfate
  Arms: Soy protein concentrate meat analog
Other: soy protein concentrate-meat analog_dephytinization — Baked dephytinized_Meat analogs-soy protein concentrate containing 58Fe as ferrous sulfate
  Arms: Soy protein concentrate meat analog without phytic acid
Other: pork meat — Meals made with minced pork meat labelled with 57Fe.
  Arms: minced pork meat

SUMMARY:
Consumption of less meat and more plant-based protein can greatly reduce the negative impact of food production on the environment. Studies show that vegan diets can decrease greenhouse gas emissions, land use, and water. However, it is important to consider the nutritional value of alternatives, as meat is a key source of nutrients like iron. Iron deficiency anemia (IDA) is estimated to be the top 5 leading causes of years lived with disability burden globally and the first cause in women. Nutritional iron deficiency anemia is often caused by low iron content and low dietary iron bioavailability. As meat, fish, and poultry are excellent sources of bioavailable iron, shifting or maintaining a predominantly plant-based diet can increase the risk of iron deficiency (ID).

Phytic acid, the main phosphorus storage compound in plants, can hinder iron absorption and other divalent minerals. Phytase is an enzyme that breaks down phytic acid, which lessens its ability to bind with minerals like iron. This enzyme is present in various plant tissues, with particularly high amounts found in wheat and rye.

There is limited clinical evidence regarding iron absorption from plant-based meat. Thus, it is important to measure iron absorption from plant-based foods before and after treatment to remove phytic acid (dephytinization).

The aim of this study is to determine the effect of phytic acid reduction on iron absorption. FIA of the soy protein concentrates meat analog with phytic acid will be compared with FIA from soy protein concentrate with dephytinization. In addition, this study will assess the FIA in a pork meat meal and will compare it to the FIA from the dephytinized meat analog.

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess the iron absorption from plant-based protein with and without the reduction of phytic acid. This study is a randomized control trial, cross-over where each participant acts as their own control.

Participants will be asked to consume test meals prepared from soy with and without dephytinization and test meals based on minced pork meat, that contains isotopic iron (57Fe and 58Fe) as ferrous sulfate. After 14 days of the test meal administration, participants will be given blood samples to access the isotopic iron enrichment in blood.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 18-45 y old
* Plasma ferritin < 30 microgram/L
* BMI 18.5-25.0
* Weight < 65 kg
* Signed informed consent

Exclusion Criteria:

* Anemic (Hb < 12 g/dL)
* Inflammation (CRP > 5 mg/L)
* Chronic digestive, renal and/or metabolic disease
* Chronic medications (except for oral contraceptives)
* Use of vitamin, mineral, and pre-and/or probiotic supplements in the previous 2 weeks and during the study
* Blood transfusion, blood donation, or significant blood loss (> 400 ml) over the past 4 months
* Difficulty with blood withdrawal
* Antibiotic treatment in the 4 weeks preceding the start of the study and during the study
* Pregnancy (tested in serum at screening) or intention to become pregnant during the course of the study
* Lactation
* Earlier participation in a study using stable isotopes or participation in any clinical study within the last 30 days
* Participants who cannot be expected to comply with the study protocol (e.g. not available on certain study appointments)
* Inability to understand the information sheet and the informed consent form due to cognitive or language reasons
* Smoking
* celiac disease or gluten intolerance
* Vegetarian or vegan dietary regimen

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women are vulnerable to developing iron deficiency. Thus, this study aims to study in female population according to sex.
Enrollment: 19 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | Baseline, 14 days after test meal administration
  The fraction of absorbed iron from isotopic iron contained in the test meal. This fractional iron absorption will be measured from blood sample after 14 days from test meal administration

SECONDARY OUTCOMES:
Iron status | Baseline, 14 days after test meal administration
  Hemoglobin (Hb), plasma ferritin (PF), and serum soluble transferrin receptor (sTfR)
Inflammatory status | Baseline, 14 days after test meal administration
  Alpha-1-acid glycoprotein (AGP), C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, Ph.D, Principal Investigator — FFHS
Locations (1):
- Fernfachhochschule Schweiz (FFHS) - Campus Gleisarena, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No